CLINICAL TRIAL: NCT04374929
Title: Subcostal Temporary Extracardiac Pacing II (STEP II) Study
Brief Title: Subcostal Temporary Extracardiac Pacing II Study
Acronym: STEP II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AtaCor Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DOC-10084
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Conduction Defect
Keywords: Temporary; Ventricular; Pacing
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Negative Pressure Wound Therapy (Active Comparator)
  Interventions: Device: StealthTrac Temporary Pacing Lead Plus Negative Pressure Wound Therapy
- Anti-Inflammatory Glucocorticoid (Active Comparator)
  Interventions: Device: StealthTrac Temporary Pacing Lead Plus Anti-Inflammatory Glucocorticoid
- Increased Electrode Spacing (Active Comparator)
  Interventions: Device: Two StealthTrac Temporary Pacing Leads (Increased Electrode Spacing)
- Control (Other)
  Interventions: Device: StealthTrac Lead Only (Control)

INTERVENTIONS:
Device: StealthTrac Temporary Pacing Lead Plus Negative Pressure Wound Therapy — Following fixation of the StealthTrac Lead, Negative Pressure Wound Therapy is applied over the incision site.
  Arms: Negative Pressure Wound Therapy
Device: StealthTrac Temporary Pacing Lead Plus Anti-Inflammatory Glucocorticoid — • Methylprednisolone 125 mg administered over 30 minutes beginning at least 30 minutes prior to the incision and StealthTrac Lead insertion procedure. This intravenous dose can be repeated every 8 hours on day one of the insertion from 1-3 doses depending on the patient's ability to take oral medications. It can be administered daily thereafter until the patient is able to take oral dosing. In normal circumstances, post op day 2, commence oral glucocorticoid (see below for recommended oral dosing).
  Oral (PO) glucocorticoid preparations and dosing:
  * Prednisone 40-60 mg orally daily based on BMI category. BMI categories: Low (<18); Medium (18-30); High (>30). Low and medium are assigned 40 mg daily. High BMI is assigned 60 mg daily dose. This while the StealthTrac lead remains in place.
  * Methylprednisolone 16-32 mg daily based on BMI (low, medium and high) while the StealthTrac Lead remains in place.
  Arms: Anti-Inflammatory Glucocorticoid
Device: Two StealthTrac Temporary Pacing Leads (Increased Electrode Spacing) — Once the first StealthTrac Lead is placed using the procedure described in the AtaCor Temporary Pacing System Instructions for Use (DOC-10085), load a second StealthTrac Lead into the same MACH I Delivery Tool, unless it was damaged during insertion of the first StealthTrac Lead, in which case a new MACH I Delivery Tool should be used.
  Insert the second StealthTrac Lead through (1) a different intercostal muscle path within the same intercostal space or (2) within an adjacent intercostal space. Increased electrode spacing is achieved by pacing between the leads.
  Arms: Increased Electrode Spacing
Device: StealthTrac Lead Only (Control) — A single StealthTrac Lead is placed with no additional treatment.
  Arms: Control

SUMMARY:
Up to 12 subjects will be enrolled (up to 8 undergoing an AtaCor Temporary Pacing System procedure) in order to evaluate initial safety and performance of the AtaCor Temporary Pacing System when used with three (3) strategies for stabilizing AtaCor Temporary Pacing System electrical measurements over a two (2) to seven (7) day period. The three treatments are (1) Negative Pressure Wound Therapy, (2) Anti-Inflammatory Glucocorticoid and (3) increased electrode spacing. A control arm with no additional treatment is also included. Safety will be evaluated through analysis of all Adverse Events. Performance will be evaluated through (1) the incidence of successful StealthTrac Lead placement using the MACH I Delivery Tool, (2) electrical performance measurements, such as pacing capture thresholds, sensed R-wave amplitudes, pacing impedance and skeletal muscle stimulation. Appropriate sensing and pacing capture will be ascertained from ECG Holter Monitor recordings during periods of in-hospital ambulation.

DETAILED DESCRIPTION:
Enrolled Subjects will have both a market-released transvenous pacing lead and investigational StealthTrac Temporary Pacing Lead placed and evaluated. Following StealthTrac Lead insertion, each subject will receive (1) one of three (3) study treatments intended to stabilize pacing capture thresholds and pacing impedance over time or receive no treatment. The three treatments are (1) Negative Pressure Wound Therapy, (2) Anti-Inflammatory Glucocorticoid and (3) increased electrode spacing achieved by the use of two inserted StealthTrac Leads. During the placement procedure, diagnostic echocardiograms will be performed to detect any new pericardial effusions. Once inserted, the StealthTrac Lead will be used to deliver high rate pacing (160 to 220 BPM) in clinically appropriate Subjects, to demonstrate suitability for use in transcatheter procedures that require brief periods of temporary pacing. Lead positions will be documented using fluoroscopic images before the Subject leaves the procedure room. On the following two days after the procedure, electrical performance will be evaluated in multiple postures and appropriate pacing and sensing will be confirmed during activity using ECG Holter monitor recordings. Subjects will also be asked patient-centric questions about their experience with the StealthTrac Lead throughout the study period. Evaluations will continue for a maximum of seven (7) days after the index procedure. Prior to StealthTrac Lead removal, an X-Ray will be taken to document the final lead position. A final follow-up will be performed 25-30 days after removal to identify any latent adverse events before the Subject exits the study.

ELIGIBILITY:
Inclusion Criteria:

1. Indicated for closed-chest cardiac invasive procedure that does not require full systemic anticoagulation during the procedure.

   Examples of such procedures include: transcatheter valve replacement, balloon valvuloplasty, implantable cardioverter-defibrillator (ICD) implantation, permanent pacemaker implantation and pacing lead extractions/revisions.
2. Physically and mentally capable of providing informed consent and at least 18 years of age or of legal age to provide consent as required by local and national requirements.

Exclusion Criteria:

1. History of a prior sternotomy (median or partial);
2. History of prior surgery with disruption of the lung, pericardium or connective tissue between the sternum and pericardium;
3. History of significant anatomic derangement of or within the thorax (e.g., pectus excavatum, significant scoliosis), prior chest radiation therapy or other reasons which may cause pericardial adhesions or complicate the AtaCor Temporary Pacing System insertion procedure;
4. History of pericardial disease, pericarditis or mediastinitis;
5. History of chronic obstructive pulmonary disease (COPD);
6. NYHA functional classification IV at the time of enrollment;
7. History of congenital heart disease;
8. Patients with circumstances that prevent data collection or follow-up;
9. BMI > 35 kg/m2;
10. Contraindication to glucocorticoid medication;
11. History of allergies to any study devices; and
12. Participation in any concurrent study without prior, written approval from the Sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Safety Outcome: Number of Subjects Experiencing an Adverse Device Effect | 30 days
  Number of Subjects Experiencing an Adverse Device Effect
Performance Outcome | Up to 7 days post insertion
  Mean Pacing Capture Threshold (V)
Performance Outcome | Up to 7 days post insertion
  Mean Pacing Impedance (Ohms)
Performance Outcome | Up to 7 days post insertion
  Mean R-Wave Amplitude (mV)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Burke, D.O., Principal Investigator — AtaCor Medical; Adrian Ebner, M.D., Principal Investigator — Sanatorio Italiano
Locations (2):
- Christchurch Hospital, Christchurch, New Zealand
- Sanatorio Italiano, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: No